CLINICAL TRIAL: NCT01431963
Title: A Multi-center, Uncontrolled, Open-label, Evaluation of Lamotrigine Monotherapy in Newly Diagnosed Epilepsy or Recurrent Epilepsy (Currently Untreated)
Brief Title: Clinical Study of Lamotrigine to Treat Newly Diagnosed Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115376
Record Dates: First submitted 2011-09-01; First posted 2011-09-12 (Estimated); Results first posted 2013-12-03 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-08

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lamotrigine (Experimental): No comparison.
  Interventions: Drug: Lamictal

INTERVENTIONS:
Drug: Lamictal — No comparison.

SUMMARY:
This is a multi-center, uncontrolled, open-label study conducted in Japan and South Korea to evaluate the efficacy and safety of lamotrigine monotherapy in subjects with newly diagnosed epilepsy and those with recurrent epilepsy (currently untreated).

The study is composed of baseline, escalation phase, maintenance phase, taper phase and post study examination. During the escalation phase, the investigational product is administered orally at 25 mg/day for 2 weeks, then 50 mg/day for 2 weeks and finally 100 mg/day for 2 weeks. During the maintenance phase, 200 mg/day is administered orally for 24 weeks. However, the dose can be decreased to 100 mg/day if there are safety concerns. Also, if it is confirmed that the seizures cannot be controlled at the dose of 200 mg/day, the dose can be gradually increased up to 400 mg/day by 50-100 mg/day at intervals of at least 1 week. As a rule, lamotrigine should be administered once daily (in the evening), but the dose exceeding 200 mg/day can be administered in two divided doses (in the morning and evening). After the completion of maintenance phase, Japanese subjects who have responded to lamotrigine without tolerability issues are eligible to enter an extension phase of the study if indicated, until either approval of this indication (monotherapy in epilepsy) or after 24 months after LSLV (Last Subject's Last Visit) of the maintenance phase, whichever is sooner.

ELIGIBILITY:
Inclusion Criteria:

1. Target disease: Subjects with newly diagnosed epilepsy or recurrent epilepsy which is untreated, having the following seizure types as classified by the International Classification of Seizures.

   * Partial seizures (with or without secondarily generalisation)
   * Generalized tonic-clonic seizures without focal onset, with or without myoclonus but without other generalized seizure type(s).
2. Subjects have a confident diagnosis of epilepsy uncomplicated by pseudoseizures (psychogenic nonepileptic seizures).
3. Subjects have had at least 2 seizures in the previous 6 months with at least 1 seizure in the previous 3 months.
4. Age: ≥16 years (at the time of obtaining consent)
5. Outpatients
6. Subjects are able to write a seizure diary.
7. Subjects understand and sign written informed consent. If a subject is under 20 years at the time of obtaining consent, a subject and a legally acceptable representative (e.g., a parent or a custodian) sign written consent to participate in this study.
8. Gender: Male or female If female, and of childbearing potential, be using an acceptable form of birth control.
9. QTc<450 millisecond (msec) or <480msec for subjects with Bundle Branch Block - values based on either single ECG values or triplicate ECG averaged QTc values obtained over a brief recording period.
10. Subjects are able to comply with dosing of investigational products and all study procedures.

Exclusion Criteria:

1. Subjects having seizure types other than partial seizure or generalized tonic clonic seizures with or without myoclonus. Subjects having status epilepticus within the 6 months prior to the start of study treatment.
2. Subjects with a history of treatment with AEDs (≥2 weeks) during 6 months before the start of treatment with the investigational product.
3. Subjects with a history of treatment with lamotrigine.
4. Subjects with a history of rash associated with other AED treatment.
5. Subjects with a history of substance (including alcohol and drugs) dependence within 12 months before the start of investigational product or abuse within 1 month before the start of investigational product according to DSM-IV-TR.
6. Subjects with an acute or chronic illness likely to impair drug absorption, distribution, metabolism or excretion or with any unstable physical symptoms likely to require hospitalization during participation in the study.
7. Subjects with a severe psychiatric disorder which affects the procedure of study or drug assessment.
8. Subjects with an acute or progressive neurological disorder or an organic disease.
9. Subjects with any clinically significant chronic cardiac, renal, or hepatic medical condition. Any patient with these conditions are excluded from the study even if these conditions are being controlled with chronic therapy.
10. Subjects with an unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, oesophageal or gastric varices or persistent jaundice), cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
11. Female subjects who are pregnant or lactating, who may be pregnant, or who plan for pregnancy during the study.
12. Subjects taking inducers of lamotrigine glucuronidation (i.e., rifampicin, lopinavir/ritonavir), atazanavir/ritonavir, risperidone, oral contraceptives or hormone drug which includes estrogen.
13. Subjects having participated in other clinical study within 3 months before the start of investigational product.
14. Subjects who have active suicidal plan/intent or have had active suicidal thoughts in the past 3 months before the start of investigational product or who have history of suicide attempt in the last 1 year before the start of investigational product or more than 1 lifetime suicide attempt.
15. Subjects whom the investigator or subinvestigator considers ineligible for the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-09; Primary Completion 2013-03 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- Japan (10):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Nara
  - GSK Investigational Site, Niigata
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Shizuoka
- GSK Investigational Site, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 115376 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115376 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115376 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115376 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115376 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 70 participants were enrolled; 3 participants were screened but withdrew from the study before prescription of the first investigational product (67), and only 65 of the participants received at least one dose of the investigational product which comprised the safety population.
Pre-assignment Details: The study consisted of a 6-week Escalation Phase, a 24-week Maintenance Phase (MP), a >=2-week Taper Phase, and a post-study examination conducted within 1-4 weeks after the last dose of lamotrigine. In Japan only, the Extension Phase was conducted until either approval for this indication or after 24 months after Last Subject Last Visit in the MP.
Groups:
- Lamotrigine: In the EP, lamotrigine 25 milligrams per day (mg/day) was orally administered once daily (QD; in the evening [PM]) as the initial dose from Week (W) 1 to W2. As a fixed dose escalation, lamotrigine 50 mg/day was orally administered QD (in the PM) from W3 to W4; 100 mg/day was administered from W5 to W6. In the MP, lamotrigine 200 mg/day was orally administered QD (in the PM) from W7 to W30. The dose could have been decreased to 100 mg/day per safety concerns. Per investigator discretion, the investigational product was discontinued if safety concerns remained. If the 200 mg/day dose did not control seizures, the dose could have been increased up to 400 mg/day by 50-100 mg/day at >=1-week intervals. A dose >200 mg/day could have been administered in 2 divided doses (in the morning and PM). In the ExP, lamotrigine was administered at 100-400 mg/day based on seizure status/safety. If a dose <100 or >400 mg/day was judged to be necessary, the participant was withdrawn from the study.
Period: Overall Study
Arm/Group | Lamotrigine
Started | 67
Begin Escalation Phase (EP; 6 Weeks) | 67
Received Treatment | 65
Complete EP (6 Weeks) | 52
Begin Maintenance Phase (MP; 24 Weeks) | 52
Complete MP (24 Weeks) | 42
Begin Extension Phase (ExP; gt= 24weeks) | 19 (Only Japanese participants in ExP,lamotrigine monotherapy was available in Korea. (>=24weeks))
Complete ExP (gt= 24 Weeks) | 19 ((>=24 weeks); gt= abbreviation for greater than or equal to)
Completed | 32
Not Completed | 35
Not completed — Adverse Event | 18
Not completed — Lack of Efficacy | 7
Not completed — Protocol Violation | 1
Not completed — Protocol-defined Stopping Criteria | 2
Not completed — Physician Decision | 4
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Baseline data were collected in members of the Safety Population, comprised of all participants who had taken at least one dose of investigational product.
Arm/Group | Lamotrigine
Number analyzed (Participants) | 65
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline data were collected in members of the Safety Population, comprised of all participants who had taken at least one dose of investigational product.
  Years | 37.3 (20.20)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline data were collected in members of the Safety Population, comprised of all participants who had taken at least one dose of investigational product.
  Participants
    Female | 26
    Male | 39
Race/Ethnicity, Customized [Number; unit: participants] — Baseline data were collected in members of the Safety Population, comprised of all participants who had taken at least one dose of investigational product.
  participants
    Asian - East Asian Heritage | 26
    Asian - Japanese Heritage | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were Seizure Free in the Maintenance Phase (Across Seizure Types and by Seizure Type Within 6 Months Prior to the Start of the Study)
Description: Participants were considered to be seizure free if they did not report any seizures during the Maintenance Phase. Seizure types are defined as: ALL=any type of seizure; A: simple partial seizures, B: complex partial seizures; C: partial seizures evolving to secondary generation seizures; D5: tonic-clonic seizures. Simple partial seizures are seizures that affect only a small region of the brain, often the temporal lobes or hippocampi. Complex partial seizures are epileptic seizures that are associated with bilateral cerebral hemisphere involvement and cause impairment of awareness or responsiveness. Partial seizures evolving to secondary generation seizures are seizures that start as partial seizures, then spread to include the entire brain. Tonic-clonic seizures are a type of generalized seizure that affects the entire brain.
Time Frame: Weeks 7 to 30
Population: Full Analysis Set (FAS): all participants in the Safety Population (SP) who provided at least one set of efficacy data after the first dosing of investigational product. The SP is comprised of all participants who had taken at least one dose of investigational product. Only those participants available at the specified time point were analyzed.
Measure: Number; unit: participants
Arm/Group | Lamotrigine
Number analyzed (Participants) | 65
participants
  All, n=65 | 28
  A+B+C, n=55 | 22
  A+B, n=42 | 17
  C, n=33 | 23
  D5, n=10 | 8
Statistical Analysis 1: Comparison: Lamotrigine; Test type: Superiority or Other; percentage of participants = 43.1, 95% CI 2-sided [30.85 to 55.96] — The estimated value reflects the percentage of participants who were seizure free for all seizures
Statistical Analysis 2: Comparison: Lamotrigine; Test type: Superiority or Other; percentage of participants = 40.0, 95% CI 2-sided [27.02 to 54.09] — The estimated value reflects the percentage of participants who were seizure free for A+B+C seizures
Statistical Analysis 3: Comparison: Lamotrigine; Test type: Superiority or Other; percentage of participants = 40.5, 95% CI 2-sided [25.63 to 56.72] — The estimated value reflects the percentage of participants who were seizure free for A+B seizures
Statistical Analysis 4: Comparison: Lamotrigine; Test type: Superiority or Other; percentage of participants = 69.7, 95% CI 2-sided [51.29 to 84.41] — The estimated value reflects the percentage of participants who were seizure free for C seizures
Statistical Analysis 5: Comparison: Lamotrigine; Test type: Superiority or Other; percentage of participants = 80.0, 95% CI 2-sided [44.39 to 97.48] — The estimated value reflects the percentage of participants who were seizure free for D5 seizures

2. Secondary Outcome: Time to Withdrawal/Dropout From the Study (Across Seizure Types and by Seizure Type in Past 6 Months in the Escalation and Maintenance Phases)
Description: Time to withdrawal is defined as the time from the start of treatment until withdrawal from the study. Seizure types are defined as: ALL=any type of seizure; A: simple partial seizures, B: complex partial seizures; C: partial seizures evolving to secondary generation seizures; D5: tonic-clonic seizures. Simple partial seizures are seizures which affect only a small region of the brain, often the temporal lobes or hippocampi. Simple partial seizures are seizures that affect only a small region of the brain, often the temporal lobes or hippocampi. Complex partial seizures are epileptic seizures that are associated with bilateral cerebral hemisphere involvement and cause impairment of awareness or responsiveness. Partial seizures evolving to secondary generation seizures are seizures that start as partial seizures, then spread to include the entire brain. Tonic-clonic seizures are a type of generalized seizure that affects the entire brain.
Time Frame: up to Week 30
Population: FAS. Only those participants available at the specified time point were analyzed.
Measure: Mean (Standard Error); unit: Days
Arm/Group | Lamotrigine
Number analyzed (Participants) | 65
Days
  All, n=65 | 150.0 (8.99)
  A+B+C, n=55 | 148.4 (9.72)
  A+B, n=42 | 147.9 (10.72)
  C, n=33 | 168.0 (10.91)
  D5, n=10 | 14.6 (0.54)

3. Secondary Outcome: Time to the First Seizure in the Maintenance Phase (Across Seizure Types and by Seizure Type)
Description: The time to the first seizure in the Maintenance Phase is measured at the time the first seizure occurred in the Maintenance Phase. Seizure types are defined as: ALL=any type of seizure; A: simple partial seizures, B: complex partial seizures; C: partial seizures evolving to secondary generation seizures; D5: tonic-clonic seizures. Simple partial seizures are seizures that affect only a small region of the brain, often the temporal lobes or hippocampi. Complex partial seizures are epileptic seizures that are associated with bilateral cerebral hemisphere involvement and cause impairment of awareness or responsiveness. Partial seizures evolving to secondary generation seizures are seizures that start as partial seizures, then spread to include the entire brain. Tonic-clonic seizures are a type of generalized seizure that affects the entire brain.
Time Frame: Weeks 7 to 30
Population: FAS. Only those participants available at the specified time point were analyzed.
Measure: Mean (Standard Error); unit: Days
Arm/Group | Lamotrigine
Number analyzed (Participants) | 52
Days
  All, n=52 | 103.0 (9.43)
  A+B+C, n=44 | 100.4 (10.44)
  A+B, n=34 | 94.2 (12.22)
  C, n=29 | 113.3 (12.06)
  D5, n=8 | NA (NA) — No participants had D5 seizures in the Maintenance Phase (MP); thus, mean time to the first D5 seizure in the MP could not be calculated.

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from study medication start until the end of treatment (up to Week 54).
Description: SAEs and non-serious AEs were collected in members of the Safety Population, comprised of all participants who had taken at least one dose of investigational product.
Groups:
- Lamotrigine: In the EP, lamotrigine 25 mg/day was orally administered QD; in the evening(PM) as the initial dose from W1 to W2. As a fixed dose escalation, lamotrigine 50 mg/day was orally administered QD(in the PM) from W3 to W4; 100 mg/day was administered from W5 to W6. In the MP, Lamotrigine 200 mg/day was orally administered QD(PM) from W7 to W30. The dose could have been decreased to 100 mg/day per safety concerns. Per investigator discretion, the investigational product was discontinued if safety concerns remained. If the 200 mg/day dose did not control seizures, the dose could have been increased up to 400 mg/day by 50-100 mg/day at greater than or equal to 1 week intervals. A dose greater than 200 mg/day could have been administered in 2 divided doses (in the morning and PM). In the ExP, lamotrigine was administered at 100-400 mg/day based on seizure status/safety. If a dose less than 100 or greater than 400 mg/day was judged to be necessary, the participant was withdrawn from the study.
Arm/Group | Lamotrigine
Serious Adverse Events (participants affected / at risk) | 8/65
Other Adverse Events (participants affected / at risk) | 38/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lamotrigine (N=65)
Haemorrhoids (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Sick sinus syndrome (Cardiac disorders) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Epilepsy (Nervous system disorders) | 2
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1
Pulmonary contusion (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lamotrigine (N=65)
Headache (Nervous system disorders) | 14
Dizziness (Nervous system disorders) | 4
Nasopharyngitis (Infections and infestations) | 15
Rash (Skin and subcutaneous tissue disorders) | 8
Nausea (Gastrointestinal disorders) | 6
Drug eruption (Skin and subcutaneous tissue disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 4
Insomnia (Psychiatric disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.